CLINICAL TRIAL: NCT01791244
Title: A Phase IV Multicenter Randomized Study to Assess the Impact of a Patient Support Program (MinSupport Plus) on Health Related Quality of Life (HRQoL) and Adherence in Patients With Relapsing Remitting Multiple Sclerosis Administered Rebif® With the RebiSmart Device
Brief Title: A Phase 4 Study to Assess the Impact of Patient Support Program on Health Related Quality of Life and Adherence in Subjects With Relapsing-Remitting Multiple Sclerosis Administered Rebif® With the RebiSmart™ Device
Acronym: RebiQoL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR 200136-560; 2012-004887-22 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; Rebif; RebiSmart; Patient support program
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Technical support for the RebiSmart™ device (Active Comparator): Subjects will be administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 microgram (mcg) subcutaneously (SC) 3 times a week in accordance to the summary of product characteristics (SPC) along with technical support for RebiSmart.
  Interventions: Drug: Rebif®
- Subject support program (MinSupport Plus) (Experimental): Subjects will be administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 mcg SC 3 times a week in accordance to the SPC along with subject support program MinSupport Plus which includes technical support for RebiSmart™ device, personal coaching regarding treatment and understanding of the disease, lifestyle guide and web support.
  Interventions: Drug: Rebif®

INTERVENTIONS:
Drug: Rebif®

SUMMARY:
This is a randomized, comparative, and multicenter study to assess the impact of a patient support program (MinSupport Plus) on health related quality of life (HRQoL) and adherence in subjects with relapsing-remitting multiple sclerosis administered Rebif® with the RebiSmart™ device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 or older
* A diagnosis of relapsing-remitting multiple sclerosis according to the revised McDonald Criteria (2010)
* Treatment with Rebif® 22 or 44 mcg subcutaneously three times a week in accordance to the Summary of product characteristics
* Rebif® administered by the RebiSmart™ device
* Provided a signed informed consent form

Exclusion Criteria:

* Has received any components, except for technical support, of MinSupport Plus prior to study entry
* Has difficulty reading and/or understanding Swedish
* Has a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* No access to computer
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Please contact the Merck Communications Service for Recruiting locations, Darmstadt, Germany
- Sweden (13):
  - Research site, Angered
  - Research site, Ängelholm
  - Research Site, Danderyd
  - Research Site, Eksjö
  - Research Site, Gävle
  - Research Site, Karlstad
  - Research Site, KS Huddinge
  - Research Site, Linköping
  - Research Site, Malmö/Lund
  - Research Site, Motala
  - Research Site, Örnsköldsvik
  - Research Site, Skövde
  - Research Site, Trollhättan

REFERENCES:
- [Derived] Landtblom AM, Guala D, Martin C, Olsson-Hau S, Haghighi S, Jansson L, Fredrikson S. RebiQoL: A randomized trial of telemedicine patient support program for health-related quality of life and adherence in people with MS treated with Rebif. PLoS One. 2019 Jul 5;14(7):e0218453. doi: 10.1371/journal.pone.0218453. eCollection 2019. PMID 31276502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 93 subjects were randomized in the study out of which 46 were randomized to MinSupport Plus (MSP) and 47 to Technical support.
Groups:
- Subject Support Program (MinSupport Plus): Subjects were administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 microgram (mcg) subcutaneously (SC) 3 times a week in accordance to the summary of product characteristics (SPC) along with subject support program MinSupport Plus which includes technical support for RebiSmart™ device, personal coaching regarding treatment and understanding of the disease, lifestyle guide and web support.
- Technical Support for the RebiSmart™ Device: Subjects were administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 mcg SC 3 times a week in accordance to the SPC along with technical support for RebiSmart.
Period: Overall Study
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Started | 46 | 47
Intent to Treat (ITT) | 38 | 39
Completed | 31 | 29
Not Completed | 15 | 18
Not completed — Adverse Event | 5 | 7
Not completed — Insufficient clinical response | 10 | 10
Not completed — Laboratory Abnormality | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires.
Groups:
- Subject Support Program (MinSupport Plus): Subjects were administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 mcg SC 3 times a week in accordance to the SPC along with subject support program MinSupport Plus which includes technical support for RebiSmart™ device, personal coaching regarding treatment and understanding of the disease, lifestyle guide and web support.
- Total: Total of all reporting groups
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Customized [Number; unit: Participants]
  Between 18 to 72 years | 38 | 39 | 77
  Greater than (>) 72 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) Psychological Score at Month 12
Description: Multiple Sclerosis Impact Scale-29 (MSIS-29) is a validated MS specific questionnaire consisting of 29 questions of which 20 addressed the physical impact component and 9 assessed the psychological impact. A combined score can be generated, or both components can be reported separately. The psychological wellbeing assessment portion of the MSIS-29 was comprised of 9 questions in which subjects rate the impact of MS on their day-to-day life from 1=no impact to 5=extreme impact. The total Psychological Score was calculated using following formula: sum of score for 9 questions - 9/0.36. The total score range ranges from 0-100 where, lower total score indicates less psychologically-related impact while a higher total score indicates greater psychologically-related impact on a subject's functioning.
Time Frame: Baseline and Month 12
Population: The ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 35.19 (24.38) | 30.48 (20.94)
  Change at Month 12 | -2.44 (19.38) | -3.04 (19.76)
Statistical Analysis 1: Comparison: Subject Support Program (MinSupport Plus) vs Technical Support for the RebiSmart™ Device; Linear mixed model, with baseline value, time, Expanded Disability Status Score (EDSS) at baseline and sex as fixed factors was used for the analysis; Test type: Superiority or Other; p = 0.9148, linear mixed model; Adjusted Mean Difference = 0.48, 95% CI 2-sided [-8.30 to 9.25]

2. Secondary Outcome: Change From Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) Psychological Score at Month 6
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 35.19 (24.38) | 30.48 (20.94)
  Change at Month 6 | -1.36 (16.82) | -1.59 (13.26)

3. Secondary Outcome: Change From Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) Total Score at Month 6 and 12
Description: Multiple Sclerosis Impact Scale-29 (MSIS-29) is a validated MS specific questionnaire consisting of 29 questions of which 20 addressed the physical impact component and 9 assessed the psychological impact. A combined score can be generated, or both components can be reported separately. The total score of the MSIS-29 was comprised of all the 29 questions in which subjects rate the impact of MS on their day-to-day life from 1=no impact to 5=extreme impact. The total Score was calculated using following formula: sum of score for 29 questions - 29/1.45. The total score range ranges from 0-100 where, lower total score indicates less psychologically-related impact while a higher total score indicates greater psychologically-related impact on a subject's functioning.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 21.81 (21.55) | 18.01 (16.61)
  Change at Month 6 | 0.56 (9.35) | 0.14 (11.19)
  Change at Month 12 | 1.00 (11.34) | 0.00 (10.45)

4. Secondary Outcome: Change From Baseline in Euro Quality of Life Questionnaire With 5 Questions Alternatives (EQ5D-5L) Summary Score at Month 6 and 12
Description: Quality of life was assessed using the EQ5D-5L score, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension comprises 5 levels with corresponding numeric scores ranging from 1 (no problems) through 5 (extreme problems) in which 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. A unique EQ5D-5L health state was defined by combining the numeric level scores for each of the 5 dimensions and the total score ranges from 5 to 25. An increase in the EQ5D-5L total score indicates worsening.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 8.84 (3.37) | 8.03 (2.30)
  Change at Month 6 | 0.18 (2.17) | 0.10 (1.76)
  Change at Month 12 | 0.05 (2.51) | -0.08 (1.86)

5. Secondary Outcome: Change From Baseline in Euro Quality of Life Questionnaire With 5 Questions Alternatives (EQ5D-5L) Visual Analogue Scale (VAS) Scale at Month 6 and 12
Description: EQ-5D-5L VAS was used to record a subject's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patient Support Program (MinSupport Plus): Subjects were administered Rebif® by the RebiSmart™ device at a dose of either 22 or 44 mcg SC 3 times a week in accordance to the SPC along with subject support program MinSupport Plus which includes technical support for RebiSmart™ device, personal coaching regarding treatment and understanding of the disease, lifestyle guide and web support.
Arm/Group | Patient Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 71.18 (20.70) | 71.49 (16.61)
  Change at Month 6 | -0.71 (11.36) | -3.38 (19.35)
  Change at Month 12 | -0.84 (16.07) | -2.31 (20.60)

6. Secondary Outcome: Percentage of Subjects With Treatment Adherence at Month 6 and 12
Description: According to the World Health Organisation (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term). Percentage of subjects with <10% missed injections (measured with the software RDS 2.0) during 6 and 12 months were reported.
Time Frame: Month 6 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of Subjects
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
Percentage of Subjects
  At Month 6 | 71.05 | 64.10
  At Month 12 | 65.79 | 53.85

7. Secondary Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Score at Month 6 and 12
Description: Fatigue Severity Scale (FSS) is a method of evaluating fatigue in multiple sclerosis and is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. The Fatigue Severity Scale is a 9-item questionnaire developed to assess the level of fatigue due to neurological disease, were each assessed on a 1-7 scale (1= no fatigue and 7= severe fatigue). The total score was calculated as the average of individual 9-items and ranged from 1 to 7 with a higher value indicating greater impairment due to fatigue.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 3.93 (1.75) | 3.98 (1.72)
  Change at Month 6 | 0.15 (0.79) | 0.05 (0.81)
  Change at Month 12 | 0.13 (0.89) | 0.08 (1.09)

8. Secondary Outcome: Change From Baseline in Modified Fatigue Impact Scale Score at Month 6 and 12
Description: The Modified Fatigue Impact Scale is a list of 21 statements describing how fatigue may affect a person's functioning. Answers ranging from 0 (Never) to 4 (Almost always). A total score ranged from a possible 0 (no fatigue impact) to 84 (almost always impacted by fatigue). A lower total score indicates less fatigue-related impact while a higher total score indicates greater fatigue-related impact on a subject's functioning.
Time Frame: Baseline, Month 6 and 12
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires.. Here, "Overall Number of subjects analyzed" signifies those subjects who were evaluable for this outcome Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 37 | 36
units on a scale
  Baseline | 29.74 (20.50) | 31.08 (19.08)
  Change at Month 6 | 3.89 (10.81) | 2.27 (9.78)
  Change at Month 12 | 3.75 (10.43) | 1.78 (10.65)

9. Secondary Outcome: Change From Baseline in Modified Fatigue Impact Scale Index at Month 6 and 12
Description: The Modified Fatigue Impact Index assesses fatigue- severity, distress, or degree of interference. Modified Fatigue Impact Scale Index was expressed in terms of percentage and ranged from 0% (no fatigue) to 100% (almost always impacted by fatigue).
Time Frame: Baseline, Month 6 and 12
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires. Here, "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome Measure.
Measure: Mean (Standard Deviation); unit: Percentage of fatigue
Arm/Group | Patient Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 37 | 36
Percentage of fatigue
  Baseline | 35.40 (24.41) | 37.00 (22.72)
  Change at Month 6 | 4.63 (12.87) | 2.71 (11.64)
  Change at Month 12 | 4.47 (12.42) | 2.12 (12.68)

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Month 6 and 12
Description: Hospital Anxiety and Depression Scale (HADS) was used to measure depression and anxiety in patients. The scale was limited to 14 questions, a practical tool for identifying and quantifying the two most common forms psychological disturbances in medical subjects. 7 of the items relate to anxiety and 7 relate to depression. Each item on the questionnaire was scored from 0-3 giving a total score between 0 and 21 for either anxiety or depression where higher score indicates more anxiety/depression.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline (Anxiety Score) | 6.13 (4.14) | 5.62 (3.21)
  Change at Month 6 (Anxiety Score) | -0.21 (2.92) | -0.56 (2.78)
  Change at Month 12 (Anxiety Score) | -0.42 (3.48) | -0.18 (3.26)
  Baseline (Depression Score) | 4.26 (3.49) | 3.72 (2.77)
  Change at Month 6 (Depression Score) | 0.61 (2.43) | 0.46 (2.85)
  Change at Month 12 (Depression Score) | 0.42 (3.61) | 0.74 (3.14)

11. Secondary Outcome: Number of Subjects With Working Ability at Month 12
Description: Working ability was assessed by measuring the number of subjects for the following categories: 1) Subjects with full sickness/disability pension, 2) Subjects who were employed or had their own business, 3) Subjects who were retired, 4) Subjects who were studying, 5) None of the above.
Time Frame: Month 12
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires. Here, "Overall Number of subjects analyzed" signifies those subjects who were evaluable for this outcome Measure.
Measure: Number; unit: Subjects
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 32 | 35
Subjects
  Subjects with full sickness/disability pension | 4 | 5
  Subjects who were employed or had own business | 22 | 25
  Subject who were retired | 2 | 2
  Subject who were studying | 3 | 2
  None of the above | 1 | 1

12. Secondary Outcome: Percentage of Subjects With Adverse Events (AE) up to Month 12
Description: AE was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment Emergent Adverse Events (TEAEs) include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Month 12
Population: The Safety Population included all subjects who were randomized and received at least 1 dose of trial treatment.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 46 | 47
Percentage of Subjects | 45.7 | 61.7

13. Secondary Outcome: Number of Subjects With Response Based on Lifestyle Questionnaire for (MinSupport Plus) at Month 6 and 12
Description: Lifestyle Questionnaire was used to assess the quality of life for subjects based on following parameters: Stress, Alcohol, Cost, Physical Aspect, Sleep, Activity and Smoking. Subjects provided their responses on the basis of three color codes: Green, Orange and Red, where Green refers to - no problem; Orange refers to - some problem and red refers to - definite/debilitating problem.
Time Frame: Month 6 and 12
Population: ITT population was used. Here, "Overall Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome Measure and "n" signifies those subjects who were evaluable for specified time points, respectively.
Measure: Number; unit: Subjects
Arm/Group | Subject Support Program (MinSupport Plus)
Number analyzed (Participants) | 32
Subjects
  Month 6: Stress: Green; n= 30 | 2
  Month 6: Stress: Orange; n= 30 | 3
  Month 6: Stress: Red; n= 30 | 3
  Month 12: Stress: Green; n= 31 | 3
  Month 12: Stress: Orange; n= 31 | 2
  Month 12: Stress: Red; n= 31 | 2
  Month 6: Alcohol: Green; n= 30 | 7
  Month 6: Alcohol: Orange; n= 30 | 1
  Month 6: Alcohol: Red; n= 30 | 1
  Month 12: Alcohol: Green; n= 32 | 6
  Month 12: Alcohol: Orange; n= 32 | 6
  Month 12: Alcohol: Red; n= 32 | 6
  Month 6: Cost: Green; n= 30 | 4
  Month 6: Cost: Orange; n= 30 | 4
  Month 6: Cost: Red; n= 30 | 4
  Month 12: Cost: Green; n= 32 | 3
  Month 12: Cost: Orange; n= 32 | 3
  Month 12: Cost: Red; n= 32 | 3
  Month 6: Physical: Green; n= 30 | 5
  Month 6: Physical: Orange; n= 30 | 2
  Month 6: Physical: Red; n= 30 | 1
  Month 12: Physical: Green; n= 32 | 5
  Month 12: Physical: Orange; n= 32 | 1
  Month 12: Physical: Red; n= 32 | 1
  Month 6: Activity: Green; n= 30 | 5
  Month 6: Activity: Orange; n= 30 | 2
  Month 6: Activity: Red; n= 30 | 1
  Month 12: Activity: Green; n= 32 | 5
  Month 12: Activity: Orange; n= 32 | 1
  Month 12: Activity: Red; n= 32 | 1
  Month 6: Sleep: Green; n= 30 | 3
  Month 6: Sleep: Orange; n= 30 | 4
  Month 6: Sleep: Red; n= 30 | 1
  Month 12: Sleep: Green; n= 32 | 3
  Month 12: Sleep: Orange; n= 32 | 2
  Month 12: Sleep: Red; n= 32 | 1
  Month 6: Smoking: Green; n= 31 | 5
  Month 6: Smoking: Orange; n= 31 | 1
  Month 6: Smoking: Red; n= 31 | 1
  Month 12: Smoking: Green; n= 32 | 5
  Month 12: Smoking: Orange; n= 32 | 1
  Month 12: Smoking: Red; n= 32 | 1

14. Secondary Outcome: Number of Subjects With Response Based on Subject Satisfaction Questionnaire at Month 12
Description: The subject satisfaction questionnaire was defined as satisfaction with overall treatment and support from health care providers during the last 12 months. Subjects were asked to rate their satisfaction by choosing either "Very discontented, discontented, contented or Very contented".
Time Frame: Month 12
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 30 | 33
Subjects
  Very discontented | 1 | 2
  Discontented | 6 | 5
  Contented | 13 | 11
  Very contented | 10 | 15

15. Secondary Outcome: Number of Subjects With Response Based on Health Care Personnel Satisfaction Questionnaire at Month 12
Description: The subject satisfaction questionnaire was defined as satisfaction with overall treatment and support from health care providers during the last 12 months. Subjects were asked to rate their satisfaction by choosing either "Very unsatisfied, unsatisfied, satisfied or very satisfied".
Time Frame: Month 12
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires. Here, "Overall Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: Subjects
Arm/Group | Subject Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Number analyzed (Participants) | 18 | 13
Subjects
  Very unsatisfied | 0 | 1
  Unsatisfied | 2 | 0
  Satisfied | 10 | 9
  Very satisfied | 6 | 3

16. Secondary Outcome: Number of Subjects With Lifestyle Goals for MinSupport Plus at Month 12
Description: Subjects defined up to 4 personal lifestyle goals during the first study week. Subjects completed the following questions related to lifestyle goals achieved during this study: 1. Was the goal achieved? (Yes/No) 2. If yes, better than expected or achieved as expected? 3. If better than expected, a lot or a little better than expected? 4. If no, a little or a lot less than expected?
Time Frame: Month 12
Population: ITT population included all subjects randomized into the trial and have completed at least 1 post-baseline assessment of the questionnaires. Here, "n" signifies subjects who were evaluable for the specific goal in this outcome measure.
Measure: Number; unit: Subjects
Arm/Group | Subject Support Program (MinSupport Plus)
Number analyzed (Participants) | 38
Subjects
  Goal 1(G1) : Goal Achieved; n= 38 | 18
  G1: Goal not Achieved; n= 38 | 4
  G1: Missing; n= 38 | 16
  G1 Achieved: Better than Expected; n= 18 | 5
  G1 Achieved: As Expected; n= 18 | 10
  G1 Achieved: Missing; n= 18 | 3
  G1Acheived:Better than Expected:Little Better;n= 5 | 4
  G1Achieved:Better than expected:Lot better; n= 5 | 0
  G1Achieved:Better than Expected: Missing; n= 5 | 1
  G1 not Achieved: Little Less; n= 4 | 1
  G1 not Achieved: Lot Less; n= 4 | 0
  G1 not Achieved: Missing; n= 4 | 3
  Goal 2 (G2): Goal Achieved; n= 38 | 3
  G2: Goal not Achieved; n= 38 | 1
  G2: Missing; n= 38 | 34
  G2 Achieved: Better than Expected; n= 3 | 2
  G2 Achieved: As Expected; n= 3 | 0
  G2 Achieved: Missing; n= 3 | 1
  G2Achieved:Better than Expected:Little Better;n= 2 | 1
  G2 Achieved: Better than Expected:Lot Better; n= 2 | 1
  G2 Achieved: Better than Expected: Missing; n= 2 | 0
  G2 not Achieved: Little Less; n= 1 | 0
  G2 not Achieved: Lot Less; n= 1 | 1
  G2 not Achieved: Missing; n= 1 | 0
  Goal 3 (G3): Goal Achieved; n= 38 | 0
  G3: Goal not Achieved; n= 38 | 1
  G3: Missing; n= 38 | 37
  G3 Achieved: As Expected; n= 0 | 0
  G3 Achieved: Better than Expected; n= 0 | 0
  G3 Achieved: Missing; n= 0 | 0
  G3 Achieved:Better than Expected:Little Better;n=0 | 0
  G3 Achieved:Better than Expected: Lot Better;n=0 | 0
  G3 Achieved: Better than Expected: Missing; n= 0 | 0
  G3 not Achieved: Little Less; n= 1 | 1
  G3 not Achieved: Lot Less; n= 1 | 0
  G3 not Achieved: Missing; n= 1 | 0
  Goal 4 (G4): Goal Achieved; n= 38 | 0
  G4: Goal not Achieved; n= 38 | 1
  G4: Missing; n= 38 | 37
  G4 Achieved: Better than Expected; n= 0 | 0
  G4 Achieved: As Expected; n= 0 | 0
  G4 Achieved: Missing; n= 0 | 0
  G4 Expected:Little Better; n= 0 | 0
  G4Achieved:Better than expected:Lot Better; n= 0 | 0
  G4 Achieved: Better than Expected: Missing; n= 0 | 0
  G4 not Achieved: Little Less; n= 1 | 0
  G4 not Achieved: Lot Less; n= 1 | 0
  G4 not Achieved: Missing; n= 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Arm/Group | Patient Support Program (MinSupport Plus) | Technical Support for the RebiSmart™ Device
Serious Adverse Events (participants affected / at risk) | 2/46 | 0/47
Other Adverse Events (participants affected / at risk) | 19/46 | 29/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Support Program (MinSupport Plus) (N=46) | Technical Support for the RebiSmart™ Device (N=47)
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Support Program (MinSupport Plus) (N=46) | Technical Support for the RebiSmart™ Device (N=47)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Retinal disorder (Eye disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Administration site pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 1
Influenza like illness (General disorders) | 2 | 2
Injection site pain (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 5
Neutralising antibodies (Investigations) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hemiparesis (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Fear of needles (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Mood swings (Psychiatric disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No